CLINICAL TRIAL: NCT04437212
Title: A Phase II Prospective, Open-label Clinical Trial of Neoadjuvant Chemoradiotherapy Combined With Perioperative Toripalimab in Patients With Locally Advanced Esophageal Squamous Cell Cancer
Brief Title: Neoadjuvant Chemoradiotherapy Combined With Perioperative Toripalimab in Locally Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renji-KY2019-174
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Advanced Esophageal Squamous Cell Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab Group (Experimental): All patients will receive radiation therapy scheme: 41.4Gy in 23 fractions over 5 weeks, concurrently with 5 cycles of paclitaxel/cisplatin (paclitaxel 45mg/m2 and cisplatin 25 mg/m2) on days 1, 8, 15, 22,29 and 2 cycles of toripalimab 240 mg every 3 weeks after chemoradiotherapy. Esophagectomy is performed 6-8 weeks after CRT completion and after operation patients received 4 cycles of toripalimab 240 mg every 3 weeks for adjuvant treatment.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Patients received toripalimab 240mg every 3 weeks 1-7 days after neoadjuvant chemoradiotherapy for 2 cycles before operation and 28-42 days after operation for 4 cycles.
  Other Names: JS-001

SUMMARY:
Neoadjuvant chemoradiotherapy (CRT) followed by surgery has become the standard treatment option for locally advanced esophageal squamous cell cancer (ESCC). However, only 20% to 40% of patients can achieve pathologic complete response (pCR) after neoadjuvant CRT with favorable prognosis and about 10% of patients have disease progression after chemoradiotherapy. How to improve the the efficacy of neoadjuvant therapy is an important clinical problem to be solved.

Immunotherapy targeting the PD-1/PD-L1 checkpoints has demonstrated promising activity in advanced EC especially in ESCC. In Keynote181 study, for patients with metastatic esophageal squamous cell carcinoma, regardless of PD-L1 expression, pembrolizumab significantly improved overall survival compared with chemotherapy. However, the efficacy and safety of immunotherapy therapy in surgery-based multidisciplinary treatment of local advanced esophageal cancer still need a lot of clinical studies to further confirm.

The aim of this study was to evaluate the efficacy and safety of the neoadjuvant chemoradiotherapy combined with perioperative toripalimab in patients with locally advanced esophageal squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years old of either gender
* Patients with histopathological confirmed resectable thoracic esophageal squamous cell carcinoma who are anti-tumor treatment-naive;
* Clinical stage of T1-4aN1-2M0 or T3-4aN0M0 according to the 8th edition of the UICC staging system;
* ECOG PS score of 0-1;
* The indexes of hematology, biochemistry and organ function meet the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L；b. neutrophil count (ANC) ≥ 1.5×109/L; c. platelets ≥ 85×109/L; d. hemoglobin ≥ 9g/dL; e. total bilirubin ≤ 14.4µmol/L; f. ALT ≤ 75U/L; g. serum creatinine ≤ 104µmol/L and creatinine clearance rate >60 mL/min;
* Women of childbearing age must undergo a pregnancy test within 7 days before enrolling in the treatment, and those who are negative can be enrolled. Patients of childbearing age and their sexual partners agree to use reliable methods of contraception before entering the study, during the study, and at least 180 days after the end of the study;
* Ability to understand the study and sign informed consent.

Exclusion Criteria:

* Patients with active infection within 2 weeks before the first use of the study drug or need to be treated with oral or intravenous antibiotics;
* A history of interstitial lung disease or non-infectious pneumonia;
* Patients whose clinician judges surgery as the first choice for the best treatment;
* A history of autoimmune diseases or abnormal immune system ;
* Patients who cannot tolerate chemoradiotherapy or surgery due to severe cardiac, lung dysfunction。
* Patients diagnosed with any other malignant tumor within 5 years before enrollment, except for malignant tumors with low risk of recurrence and risk of death, such as fully treated basal cell or squamous cell skin and carcinoma in situ of the cervix;
* Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of Toripalimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
* A history of immunodeficiency，including a positive HIV test result or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
* Women during pregnancy or lactation;
* Other situations not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response Rate (MPR) | From date of surgery to 14 days later
  No more than 10% of tumor cells were found in neoadjuvant surgical specimens.

SECONDARY OUTCOMES:
2-year disease-free survival | From date of surgery until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
2-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months
Incidence of Treatment-related Adverse Events as Assessed by CTCAE v5.0 | 60 days after the end protocol treatment
Perioperative complication rate | From date of surgery to 30 days later

CONTACTS AND LOCATIONS:
Overall Officials: Xiumei Ma, doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu X, Sun Z, Liu Q, Zhang Y, Shen L, Zhang C, Lin H, Hu B, Rong L, Chen H, Wang X, Zhao X, Bai YR, Ye Q, Ma X. Neoadjuvant chemoradiotherapy combined with sequential perioperative toripalimab in locally advanced esophageal squamous cell cancer. J Immunother Cancer. 2024 Mar 7;12(3):e008631. doi: 10.1136/jitc-2023-008631. PMID 38458635